CLINICAL TRIAL: NCT00075257
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study To Evaluate The Efficacy And Safety Of DVS-233 SR For Prevention Of Depressive Relapse In Adult Outpatients With Major Depressive Disorder
Brief Title: Study Evaluating DVS-233 SR In Adult Outpatients With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3151A1-302
Record Dates: First submitted 2004-01-07; First posted 2004-01-09 (Estimated); Last update posted 2009-08-19 (Estimated); Status verified 2009-08

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

INTERVENTIONS:
Drug: DVS-233 SR

SUMMARY:
Primary Objective: To compare the efficacy and safety of DVS-233 SR versus placebo treatment in reducing the relapse rate of depressive symptoms in subjects with major depressive disorder (MDD), and to compare the percentages of relapse in terms of time to relapse between DVS-233 SR and placebo treatment groups by using survival analysis.

Secondary Objective: To assess the response of subjects on DVS-233 SR versus placebo for the clinical global evaluation, functionality, general well-being, pain, and absence of symptoms (Hamilton Psychiatric Rating Scale for Depression, 17-item [HAM-D17] < 7).

ELIGIBILITY:
Inclusion criteria in the open-label phase:

* Outpatients
* Men and women 18 to 75 years of age, inclusive. Sexually active women participating in the study must use a medically acceptable form of contraception (Medically acceptable forms of contraception include oral contraceptives, injectable or implantable methods, intrauterine devices, or properly used barrier contraception)
* Subjects must have a primary diagnosis of MDD based on the criteria in the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV), single or recurrent episode, without psychotic features (If other allowable psychiatric diagnoses are present, MDD must be the predominant psychiatric disorder present.)

Exclusion Criteria:

* Treatment with DVS-233 SR at any time in the past
* Treatment with venlafaxine (immediate release [IR] or ER) within 90 days of study day 1
* Known hypersensitivity to venlafaxine (IR or ER)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 603 (Actual)
Dates: Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer

REFERENCES:
- [Derived] McIntyre RS, Fayyad RS, Guico-Pabia CJ, Boucher M. An Analysis of Relapse Rates and Predictors of Relapse in 2 Randomized, Placebo-Controlled Trials of Desvenlafaxine for Major Depressive Disorder. Prim Care Companion CNS Disord. 2015 Feb 26;17(1):10.4088/PCC.14m01681. doi: 10.4088/PCC.14m01681. eCollection 2015. PMID 26137355
- [Derived] Thase ME, Fayyad R, Cheng RF, Guico-Pabia CJ, Sporn J, Boucher M, Tourian KA. Effects of desvenlafaxine on blood pressure in patients treated for major depressive disorder: a pooled analysis. Curr Med Res Opin. 2015 Apr;31(4):809-20. doi: 10.1185/03007995.2015.1020365. Epub 2015 Mar 26. PMID 25758058